CLINICAL TRIAL: NCT01868022
Title: Multi-arm, Non-randomized, Open-Label Phase IB Study to Evaluate GSK3052230 in Combination With Paclitaxel and Carboplatin, or Docetaxel or as Single Agent in Subjects With Solid Malignancies and Deregulated FGF Pathway Signaling
Brief Title: Study to Evaluate GSK3052230 in Combination With Paclitaxel and Carboplatin, or Docetaxel or as Single Agent in Subjects With Solid Malignancies and Deregulated Fibroblast Growth Factor (FGF) Pathway Signaling
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117360; 2013-000354-21 (EudraCT Number)
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Neoplasms
Keywords: FGFR1; FP1039; GSK3052230; docetaxel; FGFR; carboplatin; HGS1036; squamous non-small cell lung cancer; paclitaxel
MeSH Terms: conditions — Neoplasms | interventions — FP-1039; Paclitaxel; Carboplatin; Docetaxel; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: GSK3052230 + paclitaxel/carboplatin (Experimental): Subject will receive GSK3052230 as 30-minute intravenous (i.v.) infusion once a week (Day 1, Day 8, Day 15) of each 21-day cycle + paclitaxel (constant infusion for 3 hrs) and carboplatin (constant infusion for 30 to 60 minutes) iv on Day 1 of each 21-day cycle. The number of cycles of paclitaxel/carboplatin will be limited to 4 to 6 cycles.
  Interventions: Drug: GSK3052230; Drug: paclitaxel; Drug: carboplatin
- Arm B: GSK3052230 + docetaxel (Experimental): Subject will receive GSK3052230 as 30-minute intravenous (i.v.) infusion once a week (Day 1, Day 8, Day 15) of each 21-day cycle + docetaxel as 1 hour iv infusion on Day 1 of each 21-day cycle. Subjects may continue to receive docetaxel until disease progression or as long as they are considered to derive benefit from treatment.
  Interventions: Drug: GSK3052230; Drug: docetaxel
- Arm C: GSK3052230 + pemetrexed and cisplatin (Experimental): Subject will receive GSK3052230 as 30 minute iv infusion once a week (Day 1, Day 8, Day 15) of each 21 day cycle + pemetrexed iv infusion over 10 minutes on Day 1 of each 21 day cycle followed 30 minutes later by iv Cisplatin infused over 2 hours
  Interventions: Drug: GSK3052230; Drug: pemetrexed; Drug: cisplatin

INTERVENTIONS:
Drug: GSK3052230 — A clear to opalescent, colorless to pale yellow solution for IV infusion once weekly (Day 1, Day 8, Day 15) in each 21-day cycle with unit dose strengths/dose level of 5, 10, 15, and 20 mg/kg supplied in a sterile 25 mL glass vial.
Drug: paclitaxel — paclitaxel will be from commercial stock.
  Arms: Arm A: GSK3052230 + paclitaxel/carboplatin
Drug: carboplatin — carboplatin will be from commercial stock.
  Arms: Arm A: GSK3052230 + paclitaxel/carboplatin
Drug: docetaxel — docetaxel will be from commercial stock.
  Arms: Arm B: GSK3052230 + docetaxel
Drug: pemetrexed — pemetrexed will be from commercial stock
  Arms: Arm C: GSK3052230 + pemetrexed and cisplatin
Drug: cisplatin — cisplatin will be from commercial stock
  Arms: Arm C: GSK3052230 + pemetrexed and cisplatin

SUMMARY:
This phase IB trial aims to identify anticancer activity of GSK3052230 in subjects with malignancies with abnormal dependence on FGF pathway signaling. Combination doses of GSK3052230 with standard of care chemotherapy in the first and second line or greater setting of metastatic squamous non-small cell lung cancer (NSCLC) and first line malignant pleural mesothelioma subjects will be studied in the 3+3 dose-escalation design. This will be a multi-arm, multicenter, non-randomized, parallel-group, uncontrolled, open-label Phase IB study designed to evaluate the safety, tolerability and preliminary activity of GSK3052230 in combination with paclitaxel + carboplatin (Arm A), in combination with docetaxel (Arm B), or in combination with pemetrexed + cisplatin (Arm C). Approximately 70 subjects will be enrolled in the study (approximately up to 120 may be enrolled).

ELIGIBILITY:
Inclusion Criteria

* Signed written informed consent
* Histologically or cytologically confirmed diagnosis: Arm A and B- stage IV recurrent metastatic squamous NSCLC with Fibroblast growth factor receptor 1 (FGFR1) gene amplification by central laboratory testing. Arm C- recurrent after local therapy or unresectable MPM with measurable lesions.

For specific arms the following requirements:

Arm A: Subjects who have received no prior therapy for Stage IIIB or Stage IV or recurrent metastatic disease. Note, to avoid any undue delay of initiating systemic chemotherapy for these subjects with newly diagnosed metastatic disease, it is allowed to initiate the first cycle of chemotherapy while eligibility for the study is still being determined, as long as the first dose of GSK3052230 is given no later than Cycle 2 Day 1 of chemotherapy. In addition, subjects with Stage IIIB or Stage IV disease and recurrence after previous NSCLC that has been treated with surgery and adjuvant chemotherapy or a radio- chemotherapy regimen with curative intent are eligible, provided 6 months has passed since this treatment ended.

Arm B: Subjects who have documented tumor progression (based on radiological imaging) or intolerability after receiving at least one prior line of platinum containing combination chemotherapy for Stage IIIB or Stage IV or recurrent metastatic disease. Note: Prior treatment should not include docetaxel but may have included paclitaxel.

Arm C: Subjects who have received no prior systemic therapy for MPM.

- Availability of archival tumor tissue required for assessment of deregulated FGF pathway signalling, but not limited to, FGFR1 amplification or FGF2 or FGFR1 expression. If archival tissue is not available, a fresh biopsy is required. In Arms A and B, subjects will be prospectively screened for FGFR1 gene amplification using a Fluorescence in situ hybridization (FISH) assay for the dose expansion and the MTD/MFD cohorts only. For inclusion in this study, based on the central laboratory testing, FGFR1 gene amplification must meet one of the following criteria: a ratio of FGFR1/CEN 8 of >=2; or average number of FGFR1 signals per tumor nucleus of >=6; or the percentage of tumor nuclei containing >=5 FGFR1 signals is >=50%.

In Arm C, FGF2 expression by IHC will be evaluated retrospectively in tissue samples by a central laboratory and is not a requirement for study entry.

* Measurable disease per RECIST version 1.1 (Arm A and B) and modified RECIST for Arm C.
* Male or female >=18 years of age.
* Women of childbearing potential must have a negative serum pregnancy test within 7 days of first dose of study treatment and agree to use effective contraception, from 14 days prior to the first dose of study treatment, throughout the study, and for 6 months following the last dose of chemotherapy or 4 weeks after the last dose of GSK3052230, whichever is latest. .
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception for at least 2 weeks prior to administration of the first dose of study treatment and for at least 6 months after the last dose of chemotherapy to allow for clearance of any altered sperm.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1 for Arm A and C subjects and 0-2 for Arm B.
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category
* Must have adequate organ function as defined by the following baseline values: Absolute neutrophil count >=1.5 x 10^9/Liter, Hemoglobin >=9 gram (g)/decilitre(dL), Platelets >=100 x 10^9/L, Partial thromboplastin time (PTT) <=1.25 x upper limit of normal (ULN), Albumin >=2.5 g/dL, Serum total bilirubin <=1.25 times ULN (for Arm B: <=ULN ), Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) <=2.5 times ULN (for Arm B: <=1.5 times ULN), Serum Creatinine <=1.5 x ULN, Or Measured or Calculated Creatinine Clearance >=45 mL/min (Arm A or B), >=65 mL/min (Arm C), Left ventricular ejection fraction >=50% by ECHO.

Exclusion Criteria

* For Arms A and C: Treatment with any FGFR inhibitor. For Arm B: Treatment with any anti-cancer therapy (for biological anti-cancer therapies see criteria below) during the preceding 4 weeks or within 4 half-lives of the therapy, whichever is longer.
* Receipt of any biological therapy within 6 weeks of the first dose of GSK3052230
* Unresolved toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03 (NCI CTCAE version 4.03) Grade 2 or higher from previous anti-cancer therapy, except alopecia.
* Active malignancy other than the cancer under study. Subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
* Presence of uncontrolled infection
* Prior major surgery or trauma within 28 days before first dose of study drug
* Presence of any non-healing wound, fracture, or ulcer
* Any prohibited medication(s) as described in protocol
* Conditions likely to increase the potential for abdominal perforation or fistula formation, including but not limited to:

Luminal intestinal cancers or bulky abdominal disease. Presence or history of abdominal fistula, gastrointestinal perforation, peptic ulcer disease or intra-abdominal abscess within the six months prior to the first dose of GSK3052230.

Other risk factors for perforation, such as acute diverticulitis, obstruction or previous abdominal or pelvic radiation.

* Symptomatic leptomeningeal or brain metastases or spinal cord compression Note: Subjects previously treated for these conditions are eligible if they meet both of the criteria below: (1) have had stable CNS disease for at least 4 weeks after local therapy as assessed by imaging (contrast enhanced magnetic resonance imaging [MRI] or computed tomography [CT]) prior to Day 1, and (2) are asymptomatic and off corticosteroids, or are on stable dose of corticosteroids for at least 4 weeks prior to Day 1.
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drugs (GSK3052230, docetaxel, paclitaxel, carboplatin, pemetrexed, cisplatin) and or their excipients that contraindicate their participation.
* Known human immunodeficiency virus-positive serology, acquired immunodeficiency syndrome (AIDS), or an AIDS-related illness.
* Prior organ or allogeneic stem cell transplant
* The following cardiac abnormalities:

Corrected QT (QTc) interval >=480 millisecond. History of acute coronary syndromes (including unstable angina) within the past 24 weeks Coronary angioplasty or stenting within the past 24 weeks. Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.

Abnormal cardiac valve morphology (>= Grade 2) documented by echocardiogram (subjects with Grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study).

History of known arrhythmias (except sinus arrhythmia and atrial fibrillation that is controlled) within the past 24 weeks.

* Presence or history of hemoptysis (>1/2 teaspoon of red blood) 2 weeks prior to the first dose of GSK3052230
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases or otherwise stable chronic liver disease per investigator's assessment).
* Pregnant, lactating or actively breast feeding females.
* French subjects: The French subject has participated in any study using an investigational study treatment(s) during the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-10-09 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- United States (10):
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Charleston, South Carolina
- GSK Investigational Site, Leuven, Belgium
- GSK Investigational Site, Koebenhavn Oe, Denmark
- GSK Investigational Site, Amsterdam, Netherlands
- Russia (4):
  - GSK Investigational Site, Arkhangelsk
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Vsevolozhsk
- Spain (5):
  - GSK Investigational Site, Badajoz
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Seville
- United Kingdom (3):
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, London
  - GSK Investigational Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=117360

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-randomized, parallel-group study in participants (par.) with Solid Malignancies and Deregulated Fibroblast growth factor (FGF) Pathway Signaling. Participants administered GSK3052230 in combination with paclitaxel + carboplatin (Arm A) or in combination with docetaxel (Arm B) or in combination with pemetrexed + cisplatin (Arm C).
Pre-assignment Details: Total 65 participants were enrolled in 3 Arms. In Arm A 20 participants were enrolled across 3 cohorts, Arm B 9 participants were enrolled across 3 cohorts, Arm C 36 participants were enrolled across 3 cohorts.The study was conducted at 22 centers across 7 countries from 9-Oct-2013 to 24-Oct-2017.
Groups:
- 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A: Participants in Arm A received 5 milligram per kilogram (mg/kg) GSK3052230 along with 200 mg per meter square (mg/m^2) of Paclitaxel plus Area under curve (AUC) 6 that is (i.e.) 900 mg Carboplatin
- 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A: Participants in Arm A received 10 mg/kg GSK3052230 along with 200 mg/m^2 of Paclitaxel plus AUC 6 i.e. 900 mg Carboplatin
- 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A: Participants in Arm A received 20 mg/kg GSK3052230 along with 200 mg/m^2 of Paclitaxel plus AUC 6 i.e. 900 mg Carboplatin
- 5 mg/kg GSK3052230 + Docetaxel: Arm B: Participants in Arm B received 5 mg/kg GSK3052230 along with 75 mg/m^2 Docetaxel
- 10 mg/kg GSK3052230 + Docetaxel: Arm B: Participants in Arm B received 10 mg/kg GSK3052230 along with 75 mg/m^2 Docetaxel
- 20 mg/kg GSK3052230 + Docetaxel: Arm B: Participants in Arm B received 20 mg/kg GSK3052230 along with 75 mg/m^2 Docetaxel
- 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C: Participants in Arm C received 10 mg/kg GSK3052230 along with 500 mg/m^2 Pemetrexed plus 75 mg/m^2 Cisplatin
- 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C: Participants in Arm C received 15 mg/kg GSK3052230 along with 500 mg/m^2 Pemetrexed plus 75 mg/m^2 Cisplatin
- 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C: Participants in Arm C received 20 mg/kg GSK3052230 along with 500 mg/m^2 Pemetrexed plus 75 mg/m^2 Cisplatin
Period: Overall Study
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Started | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 25 | 8
Completed | 3 | 3 | 13 | 2 | 1 | 2 | 3 | 16 | 6
Not Completed | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 9 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Study closed/terminated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Ongoing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | Total
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 25 | 8 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.0 (5.29) | 71.7 (5.03) | 65.0 (7.55) | 58.0 (8.19) | 67.0 (12.00) | 65.7 (5.77) | 72.3 (7.51) | 57.1 (13.90) | 70.9 (6.06) | 66.52 (3.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 8 | 2 | 13
  Male | 3 | 3 | 13 | 3 | 3 | 2 | 2 | 17 | 6 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Arabic/North African Heritage | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White - White/Caucasian/European Heritage | 2 | 3 | 14 | 3 | 3 | 3 | 3 | 24 | 8 | 63
  Asian - Central/South Asian Heritage | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-serious Adverse Events (AEs) and Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, protocol-specific events including drug-induced liver injury with hyperbilirubinaemia, any new primary cancers, cardiac toxicity including Left Ventricular Ejection Fraction (LVEF) changes or treatment emergent cardiac valve toxicity and treatment emergent acute anterior uveitis were categorized as SAE. Participants having non-serious AE or SAE were included in the analysis. The All Treated Subjects Population comprised of all participants who received at least one dose of study treatment.
Time Frame: Median of 28.5 weeks
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 25 | 8
Participants
  Non-serious AEs | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 24 | 8
  SAEs | 0 | 3 | 5 | 2 | 3 | 1 | 0 | 5 | 4

2. Primary Outcome: Number of Participants With Severe AEs and SAEs
Description: The severity of AEs were graded utilizing National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.3. Grade 1 represents mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 represents moderate; minimal, local or noninvasive intervention indicated. Grade 3 represents severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling. Grade 4 represents life-threatening consequences; urgent intervention indicated. Grade 5 represents death related to AE.
Time Frame: Median of 28.5 weeks
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 25 | 8
Participants
  Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 7 | 1
  Grade 3 | 1 | 1 | 8 | 2 | 2 | 0 | 1 | 17 | 4
  Grade 4 | 2 | 2 | 4 | 1 | 1 | 3 | 0 | 0 | 2
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Number of Participants Withdrew Due to AEs
Description: An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. The AEs leading to permanent discontinuation from the study has been reported.
Time Frame: Median of 28.5 weeks
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 25 | 8
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 3

4. Primary Outcome: Number of Participants With Dose Reduction
Description: Dose reduction and delays were done due to toxicity, or in the interest of participant's safety per investigator discretion. Requirement for more than 2 dose reductions resulted in permanent discontinuation of chemotherapy. Participants with dose reduction has been reported.
Time Frame: Median of 28.5 weeks
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 25 | 8
Participants | 1 | 0 | 3 | 1 | 0 | 2 | 0 | 2 | 0

5. Primary Outcome: Number of Participants With Dose Delays
Description: Dose reduction and delays were done due to toxicity, or in the interest of participant's safety per investigator discretion. Requirement for more than 2 dose reductions resulted in permanent discontinuation of chemotherapy. Participants with dose delay has been reported.
Time Frame: Median of 28.5 weeks
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 25 | 8
Participants | 0 | 2 | 4 | 2 | 1 | 0 | 2 | 12 | 1

6. Primary Outcome: Treatment Duration With GSK3052230
Description: The number of participants administered study treatment were summarized according to the duration of therapy. The extent of treatment exposure is calculated as the number of cycles administered. The duration of exposure to study treatment is calculated from first day to last day of treatment plus 1 day. Median and full range (minimum and maximum) has been reported.
Time Frame: Median of 28.5 weeks
Population: All Treated Subjects Population
Measure: Median (Full Range); unit: Cycles
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 25 | 8
Cycles | 7.0 [3 to 8] | 15.0 [5 to 20] | 8.0 [2 to 13] | 6.0 [2 to 7] | 4.0 [2 to 14] | 6.0 [3 to 8] | 6.0 [4 to 8] | 11.0 [1 to 23] | 3.0 [1 to 32]

7. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: DLT is defined as toxicities due to GSK3052230 or due to the combination of GSK3052230 with chemotherapy within Cycle 1 (first 21 days of period on study) that are unlikely to be due to another cause, such as the known effects of cytotoxics chemotherapy alone, disease progression, or accident, and protocol-specified criteria. Clinically significant toxicities that persist or occur beyond Cycle 1 that the investigator and GlaxoSmithKline (GSK) medical monitor consider dose-limiting may also be designated a DLT for the purpose of establishing Maximum tolerated dose (MTD). Number of participants with DLTs has been reported.
Time Frame: Median of 28.5 weeks
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 25 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3

8. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure was measured in a semi-supine position after 5 minutes of rest. Blood pressure was measured before start of first chemotherapy infusion and within 20 minutes before start of GSK3052230 infusion on Day 1 of every cycle and Baseline. Baseline is defined as the most recent, non-missing value prior to or on the first study GSK3052230 treatment dose date. Change from Baseline is calculated as visit value minus Baseline value. The worst-case post-Baseline values has been presented. NA indicates that data were not available as standard deviation could not be calculated for a single participant. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to Median of 28.5 weeks
Population: All Treated Subjects Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 25 | 8
Millimeters of mercury (mmHg)
  DBP, n=3, 2, 9, 3, 2, 2, 3, 21, 5: number analyzed (Participants) | 3 | 2 | 9 | 3 | 2 | 2 | 3 | 21 | 5
  DBP, n=3, 2, 9, 3, 2, 2, 3, 21, 5 | 6.3 (16.17) | 0.5 (12.02) | 2.0 (10.39) | -0.6 (3.06) | 6.0 (2.83) | 3.5 (9.19) | 2.3 (7.64) | 12.8 (8.38) | 10.6 (2.30)
  SBP, n=3, 1, 13, 2, 2, 2, 3, 21, 4: number analyzed (Participants) | 3 | 1 | 13 | 2 | 2 | 2 | 3 | 21 | 4
  SBP, n=3, 1, 13, 2, 2, 2, 3, 21, 4 | -12.3 (15.31) | -14.0 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant. | 9.6 (10.16) | 10.5 (14.85) | 17.5 (3.54) | 6.0 (22.63) | 3.0 (13.00) | 12.5 (13.21) | 18.7 (15.97)

9. Primary Outcome: Change From Baseline in Heart Rate
Description: Heart rate was measured in a semi-supine position after 5 minutes of rest. Heart rate was measured before start of first chemotherapy infusion and within 20 minutes before start of GSK3052230 infusion on Day 1 of every cycle and Baseline. Baseline is defined as the most recent, non-missing value prior to or on the first study GSK3052230 treatment dose date. Change from Baseline is calculated as visit value minus Baseline value. The worst-case post-Baseline values has been presented.
Time Frame: Baseline and up to Median of 28.5 weeks
Population: All Treated Subjects Population. Number of par. analyzed > number of par. started in the study, as these were bi-directional vital signs tests. Heart rate had both clinically significant low and high ranges and there were par. who experienced both worst case post-Baseline values.Only those par. available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Units Other Than Participants: Heart rate readings
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 25 | 7
Number analyzed (Heart rate readings) | 3 | 4 | 17 | 3 | 4 | 3 | 3 | 26 | 7
Beats per minute (bpm) | -0.3 (15.31) | 3.2 (24.74) | 8.0 (23.67) | 28.0 (42.79) | 10.5 (19.33) | 0.6 (3.06) | -5.0 (1.73) | 2.8 (20.49) | 24.4 (21.56)

10. Primary Outcome: Change From Baseline in Temperature
Description: Temperature was measured in a semi-supine position after 5 minutes of rest. Temperature was measured before start of first chemotherapy infusion and within 20 minutes before start of GSK3052230 infusion on Day 1 of every cycle and Baseline. Baseline is defined as the most recent, non-missing value prior to or on the first study GSK3052230 treatment dose date. Change from Baseline is calculated as visit value minus Baseline value. The worst-case post-Baseline values has been presented.
Time Frame: Baseline and up to Median of 28.5 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Degree Celsius
Units Other Than Participants: Temperature readings
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 14 | 2 | 3 | 3 | 3 | 25 | 8
Number analyzed (Temperature readings) | 3 | 4 | 14 | 2 | 3 | 3 | 3 | 27 | 8
Degree Celsius | -0.30 (0.361) | -0.38 (0.608) | 0.35 (0.917) | 0.10 (0.283) | 1.03 (1.795) | -0.03 (0.058) | -0.23 (0.208) | -0.16 (0.899) | 0.12 (0.742)

11. Primary Outcome: Number of Participants With Clinically Significant Findings for 12-lead Electrocardiogram (ECG)
Description: A single 12-lead ECG was performed at the specified timepoints during the study where the participant was instructed to be in semi-recumbent position for 5 minutes before obtaining the ECG. An ECG machine that automatically calculated the heart rate and measures like the PR, QRS, QT, and corrected QT intervals. Number of participants with worst-case post-Baseline abnormal clinically significant findings and abnormal not clinically significant findings in ECG results has been reported.
Time Frame: Median of 28.5 weeks
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 25 | 8
Participants
  Abnormal not clinically significant | 0 | 2 | 8 | 2 | 2 | 3 | 1 | 12 | 2
  Abnormal clinically significant | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 3

12. Primary Outcome: Number of Participants With Abnormal Echocardiogram (ECHO) Findings
Description: Echocardiography scans were obtained at given time points using an echocardiogram and the findings for left ventricular ejection fraction (LVEF) were obtained. LVEF values at end of treatment (EOT) were recorded as no change or any increase and any decrease values. Only those participants available at the specified time points were analyzed.
Time Frame: Median of 28.5 weeks
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 1 | 0 | 2 | 1 | 0 | 2 | 0 | 5 | 2
Participants
  No change or any increase | 0 |  | 1 | 0 |  | 1 |  | 2 | 2
  Any Decrease | 1 |  | 1 | 1 |  | 1 |  | 3 | 0

13. Primary Outcome: Number of Participants With Clinical Chemistry Changes From Baseline With Respect to the Normal Range
Description: Clinical chemistry parameters included potassium, sodium, chloride (Cl), total carbon dioxide (CO2), total and ionized calcium, magnesium, phosphate, albumin, glucose (fasting), Blood urea nitrogen (BUN), creatinine (Cr), uric acid, creatinine clearance, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transferase (GGT), alkaline phosphatase, Total bilirubin (T. Bil), and Direct bilirubin (D. Bil), total T3 and T4, free T4, amylase, lipase, prothrombin time, partial thromboplastin time, international normalized ratio, and fibrinogen. Baseline is defined as the most recent, non-missing value prior to or on the first study GSK3052230 treatment dose date. Change from Baseline is calculated as visit value minus Baseline value. Clinical chemistry parameters with change from Baseline with respect to normal range only has been presented. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Median of 28.5 weeks
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 25 | 8
Participants
  D.Bil, decrease to low, n=2,2,8,1,2,2,1,12,6: number analyzed (Participants) | 2 | 2 | 8 | 1 | 2 | 2 | 1 | 12 | 6
  D.Bil, decrease to low, n=2,2,8,1,2,2,1,12,6 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  D.Bil, normal or no change, n=2,2,8,1,2,2,1,12,6: number analyzed (Participants) | 2 | 2 | 8 | 1 | 2 | 2 | 1 | 12 | 6
  D.Bil, normal or no change, n=2,2,8,1,2,2,1,12,6 | 2 | 1 | 7 | 1 | 2 | 1 | 1 | 7 | 5
  D.Bil, increase to high, n=2,2,8,1,2,2,1,12,6: number analyzed (Participants) | 2 | 2 | 8 | 1 | 2 | 2 | 1 | 12 | 6
  D.Bil, increase to high, n=2,2,8,1,2,2,1,12,6 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 5 | 1
  Cl, decrease to low, n=3,3,14,3,3,3,3,25,8 | 1 | 1 | 5 | 0 | 2 | 1 | 2 | 9 | 3
  Cl, normal or no change, n=3,3,14,3,3,3,3,25,8 | 2 | 0 | 8 | 3 | 1 | 2 | 1 | 15 | 5
  Cl, increase to high, n=3,3,14,3,3,3,3,25,8 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 2
  CO2, decrease to low, n=3,3,14,3,3,3,3,25,8 | 0 | 1 | 3 | 1 | 0 | 0 | 1 | 2 | 0
  CO2, normal or no change, n=3,3,14,3,3,3,3,25,8 | 2 | 1 | 8 | 2 | 3 | 1 | 2 | 17 | 5
  CO2, increase to high, n=3,3,14,3,3,3,3,25,8 | 1 | 2 | 6 | 0 | 0 | 2 | 0 | 7 | 3
  Cr CL, decrease to low, n=3,3,9,2,1,3,3,15,4: number analyzed (Participants) | 3 | 3 | 9 | 2 | 1 | 3 | 3 | 15 | 4
  Cr CL, decrease to low, n=3,3,9,2,1,3,3,15,4 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 9 | 0
  Cr CL, normal or no change, n=3,3,9,2,1,3,3,15,4: number analyzed (Participants) | 3 | 3 | 9 | 2 | 1 | 3 | 3 | 15 | 4
  Cr CL, normal or no change, n=3,3,9,2,1,3,3,15,4 | 2 | 1 | 8 | 1 | 1 | 3 | 2 | 6 | 4
  Cr CL, increase to high, n=3,3,9,2,1,3,3,15,4: number analyzed (Participants) | 3 | 3 | 9 | 2 | 1 | 3 | 3 | 15 | 4
  Cr CL, increase to high, n=3,3,9,2,1,3,3,15,4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  T4 free, decrease to low, n=0,1,6,0,1,0,2,16,3: number analyzed (Participants) | 0 | 1 | 6 | 0 | 1 | 0 | 2 | 16 | 3
  T4 free, decrease to low, n=0,1,6,0,1,0,2,16,3 |  | 0 | 1 |  | 0 |  | 0 | 1 | 1
  T4 free, normal or no change,=0,1,6,0,1,0,2,16,3: number analyzed (Participants) | 0 | 1 | 6 | 0 | 1 | 0 | 2 | 16 | 3
  T4 free, normal or no change,=0,1,6,0,1,0,2,16,3 |  | 1 | 5 |  | 1 |  | 2 | 12 | 2
  T4 free, increase to high, n=0,1,6,0,1,0,2,16,3: number analyzed (Participants) | 0 | 1 | 6 | 0 | 1 | 0 | 2 | 16 | 3
  T4 free, increase to high, n=0,1,6,0,1,0,2,16,3 |  | 0 | 0 |  | 0 |  | 0 | 3 | 0
  T4 total, decrease to low, n=0,0,0,0,0,0,1,4,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1
  T4 total, decrease to low, n=0,0,0,0,0,0,1,4,1 |  |  |  |  |  |  | 0 | 1 | 0
  T4 total, normal or no change, n=0,0,0,0,0,0,1,4,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1
  T4 total, normal or no change, n=0,0,0,0,0,0,1,4,1 |  |  |  |  |  |  | 1 | 1 | 0
  T4 total, increase to high, n=0,0,0,0,0,0,1,4,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1
  T4 total, increase to high, n=0,0,0,0,0,0,1,4,1 |  |  |  |  |  |  | 0 | 2 | 1
  Total T3, decrease to low, n=0,1,1,0,1,0,1,6,3: number analyzed (Participants) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 6 | 3
  Total T3, decrease to low, n=0,1,1,0,1,0,1,6,3 |  | 0 | 0 |  | 0 |  | 0 | 3 | 2
  Total T3, normal or no change, n=0,1,1,0,1,0,1,6,3: number analyzed (Participants) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 6 | 3
  Total T3, normal or no change, n=0,1,1,0,1,0,1,6,3 |  | 1 | 1 |  | 1 |  | 1 | 2 | 1
  Total T3, increase to high, n=0,1,1,0,1,0,1,6,3: number analyzed (Participants) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 6 | 3
  Total T3, increase to high, n=0,1,1,0,1,0,1,6,3 |  | 0 | 0 |  | 0 |  | 0 | 1 | 0
  Urea/BUN, decrease to low, n=3,2,13,3,2,3,3,25,8: number analyzed (Participants) | 3 | 2 | 13 | 3 | 2 | 3 | 3 | 25 | 8
  Urea/BUN, decrease to low, n=3,2,13,3,2,3,3,25,8 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 1
  Urea/BUN,normal or no change,n=3,2,13,3,2,3,3,25,8: number analyzed (Participants) | 3 | 2 | 13 | 3 | 2 | 3 | 3 | 25 | 8
  Urea/BUN,normal or no change,n=3,2,13,3,2,3,3,25,8 | 2 | 2 | 8 | 1 | 2 | 2 | 1 | 11 | 3
  Urea/BUN, increase to high, n=3,2,13,3,2,3,3,25,8: number analyzed (Participants) | 3 | 2 | 13 | 3 | 2 | 3 | 3 | 25 | 8
  Urea/BUN, increase to high, n=3,2,13,3,2,3,3,25,8 | 0 | 0 | 5 | 1 | 0 | 1 | 2 | 10 | 4

14. Primary Outcome: Number of Participants With the Abnormal Urinalysis Findings
Description: Urinalysis parameters included urine protein, urine glucose, urine ketones and occult blood were assessed. Dipstick test was performed for routine urinalysis. Abnormal values such as trace, 1+, 2+, 3+, 4+, >1000, >=1000, and >10 have been reported.
Time Frame: Up to Cycle 16 (each cycle was of 21 days)
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 25 | 8
Participants
  Cycle 1 Day 1, Urine glucose, >1000 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 1, Urine glucose, 2+ | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 1, Urine glucose, trace | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 2 Day 1, Urine glucose, trace | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 4 Day 1, Urine glucose, >=1000 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1, Urine glucose, 4+ | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 1 Day 1, Urine ketones, trace | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Cycle 4 Day 1, Urine ketones, trace | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 28, Day 1, Urine ketones, trace | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 1 Day 1, Occult Blood, 1+ | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 1 Day 1, Occult Blood, 3+ | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 2 Day 1, Occult Blood, 1+ | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Cycle 2 Day 1, Occult Blood, trace | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 4 Day 1, Occult Blood, trace | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 4 Day 1, Occult Blood, 1+ | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1, Occult Blood, 2+ | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 8 Day 1, Occult Blood, 1+ | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 1 Day 1, Urine protein, 1+ | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Cycle 1 Day 1, Urine protein, trace | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0
  Cycle 2, Day 1, Urine protein, trace | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
  Cycle 2, Day 1, Urine protein, 2+ | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 4, Day 1, Urine protein, trace | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  Cycle 8, Day 1, Urine protein, trace | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  Cycle 12, Day 1, Urine protein, trace | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 16, Day 1, Urine protein, trace | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Number of Participants With Hematology Change From Baseline With Respect to the Normal Range
Description: Hematology parameters included platelet Count, red blood cell (RBC) Count, hemoglobin, absolute white blood cell (WBC) Count, absolute neutrophils (Neu), absolute lymphocytes (Lym), absolute monocytes (Mono), absolute eosinophils (Eos), absolute basophils (Baso). Baseline is defined as the most recent, non-missing value prior to or on the first study GSK3052230 treatment dose date. Change from Baseline is calculated as visit value minus Baseline value. Hematology parameters with worst-case change from Baseline with respect to normal range only has been presented. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Median of 28.5 weeks
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 25 | 8
Participants
  Baso, decrease to low, n=3,3,14,3,3,3,3,22,8: number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 22 | 8
  Baso, decrease to low, n=3,3,14,3,3,3,3,22,8 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 5 | 1
  Baso, normal or no change, n=3,3,14,3,3,3,3,22,8: number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 22 | 8
  Baso, normal or no change, n=3,3,14,3,3,3,3,22,8 | 3 | 3 | 9 | 3 | 1 | 3 | 3 | 13 | 6
  Baso, increase to high, n=3,3,14,3,3,3,3,22,8: number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 22 | 8
  Baso, increase to high, n=3,3,14,3,3,3,3,22,8 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 4 | 1
  Eos, decrease to low, n=3,3,14,3,3,3,3,24,8: number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 24 | 8
  Eos, decrease to low, n=3,3,14,3,3,3,3,24,8 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 8 | 3
  Eos, normal or no change, n=3,3,14,3,3,3,3,24,8: number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 24 | 8
  Eos, normal or no change, n=3,3,14,3,3,3,3,24,8 | 3 | 3 | 11 | 3 | 3 | 3 | 3 | 14 | 5
  Eos, increase to high, n=3,3,14,3,3,3,3,24,8: number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 3 | 3 | 24 | 8
  Eos, increase to high, n=3,3,14,3,3,3,3,24,8 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 5 | 1
  Mono, decrease to low, n=3,3,14,3,3,3,3,25,8 | 3 | 2 | 11 | 0 | 2 | 1 | 2 | 6 | 3
  Mono, normal or no change, n=3,3,14,3,3,3,3,25,8 | 1 | 0 | 4 | 2 | 0 | 0 | 2 | 12 | 3
  Mono, increase to high, n=3,3,14,3,3,3,3,25,8 | 0 | 3 | 5 | 1 | 3 | 2 | 0 | 10 | 5
  RBC, decrease to low, n=3,3,14,3,3,3,3,25,8 | 3 | 2 | 10 | 0 | 1 | 2 | 1 | 17 | 3
  RBC, normal or no change, n=3,3,14,3,3,3,3,25,8 | 0 | 1 | 4 | 3 | 2 | 1 | 2 | 9 | 4
  RBC, increase to high, n=3,3,14,3,3,3,3,25,8 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 1

16. Primary Outcome: Number of Participants With Maximum Tolerated Dose (MTD) or Maximum Feasible Dose (MFD)
Description: The MTD is defined as the highest dose level tested at which < 33 percent of participants experience a DLT. In cases when MTD is not reached dose was described as the MFD.
Time Frame: Median of 28.5 weeks
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Groups:
- 15 mg/kg GSK3052230 + Pemetrexed + Carboplatin: Arm C: Participants in Arm C received 15 mg/kg GSK3052230 along with 500 mg/m^2 Pemetrexed plus 75 mg/m^2 Cisplatin
Arm/Group | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 15 mg/kg GSK3052230 + Pemetrexed + Carboplatin: Arm C
Number analyzed (Participants) | 14 | 3 | 25
Participants | 14 | 3 | 25

17. Primary Outcome: Number of Participants With Best Response
Description: Best response defined as complete response (CR:disappearance of all target. Any pathological lymph nodes < 10 millimeter [mm] in the short axis) or partial response (PR at least a 30 percent decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters), stable disease (SD neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease) or progressive disease (PR at least a 20 percent increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started. In addition, the sum must have an absolute increase from nadir of 5 mm) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or modified RECIST. Best response as per RECIST version 1.1 for Arm A and B participants has been reported. Best response according to RECIST version 1.1 or modified RECIST for Arm C participants has been reported.
Time Frame: Median of 28.5 weeks
Population: All Evaluable Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 13 | 3 | 3 | 3 | 3 | 25 | 8
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 1 | 2 | 6 | 0 | 0 | 0 | 2 | 11 | 1
  Stable disease, discontinued | 1 | 1 | 5 | 2 | 2 | 2 | 1 | 10 | 2
  Stable disease, ongoing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Progressive disease | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1

18. Primary Outcome: Number of Participants With Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) is defined as the percentage of participants achieving a confirmed Complete response (CR) or Partial response (PR) from the start of treatment until disease progression as per RECIST version 1.1 or modified RECIST for participants in Arm C. This was determined based on Investigator assessments of response. 95% confidence intervals (CI) are calculated based on the unconditional exact method. ORR as per RECIST vesrion 1.1 for Arm A and B has been reported. ORR as per RECIST version 1.1 and modified RECIST version 1.1 for Arm C has been reported. The study population used for decision-making at the interim analyses during the dose expansion cohorts of the study arms is termed as the All Evaluable Participants Population. NA indicates 0 participants met ORR criteria therefore no dispersion.
Time Frame: Median of 28.5 weeks
Population: All Evaluable Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 13 | 3 | 3 | 3 | 3 | 25 | 8
Participants | 1 | 2 | 6 | 0 | 0 | 0 | 2 | 11 | 1

19. Secondary Outcome: Progression Free Survival (PFS) as Assessed by Investigator
Description: PFS is defined as the interval between first dose of GSK3052230 and the earliest date of disease progression or death due to any cause by investigator assessment per RECIST 1.1 (for Arm A and B participants) or modified RECIST (for Arm C participants). For participants who do not progress or die, PFS was censored at the time of last radiological scan. Participants who discontinued study with no post-treatment tumor assessment were censored at date of first dose of study drug. Mean and 95 percent CI has been reported. NA indicates that data were not available as only 1 participant had event, other two censored therefore there is no confidence interval.
Time Frame: Median of 28.5 weeks
Population: All Evaluable Subjects Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 3 | 13 | 3 | 3 | 3 | 3 | 25 | 8
Months | 4.1 [1.4 to 5.5] | NA [5.0 to NA] — NA indicates that data were not available as only 1 participant had event, other two censored therefore there is no confidence interval | 5.5 [3.7 to 6.2] | 4.6 [1.3 to 4.6] | 9.5 [NA to NA] — NA indicates that data were not available as only 1 participant had event, other two censored therefore there is no confidence interval | 5.1 [4.0 to 6.2] | 4.6 [NA to NA] — NA indicates that data were not available as only 1 participant had event, other two censored therefore there is no confidence interval | 7.4 [6.7 to 13.4] | 4.1 [0.9 to 8.3]

20. Secondary Outcome: Clearance of GSK3052230
Description: Serial blood sample were collected at an indicated time points. A nonlinear mixed effects model was used to determine clearances. The Pharmacokinetic Population (PK) consisted of all participants in the All Treated Subject Population for whom a blood sample for pharmacokinetics was obtained and analyzed. Plasma GSK3052230 concentration-time data were to be combined with data from other studies to be analyzed using a population PK approach. However, other studies with GSK3052230 were not performed and thus no population PK analyses were done.
Time Frame: Cycle(C)1 Day (D) 1 Pre-dose, End of infusion, 1 and 2 hours post-dose;C1 D8 Pre-dose,end of infusion; C2 D1 Pre-dose, End of infusion, 1 and 2 hours post-dose;C4 D1 Predose, end of infusion;C6 D1 Pre-dose, end of infusion,C12 D1 Pre-dose, end of infusion
Population: Pharmacokinetic Population
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Volume of Distribution of GSK3052230
Description: Serial blood sample were collected at an indicated time points. A nonlinear mixed effects model was used to determine volume distribution. Plasma GSK3052230 concentration-time data were to be combined with data from other studies to be analyzed using a population PK approach. However, other studies with GSK3052230 were not performed and thus no population PK analyses were done.
Time Frame: as for outcome 20
Population: Pharmacokinetic Population
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Relevant Covariates That Influence Exposure of GSK3052230
Description: Relevant covariates included parameters like age, weight and disease related covariates. Plasma GSK3052230 concentration-time data were to be combined with data from other studies to be analyzed using a population PK approach. However, other studies with GSK3052230 were not performed and thus no population PK analyses were done.
Time Frame: as for outcome 20
Population: Pharmacokinetic Population
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) in of Arm C Participants With Malignant Pleural Mesothelioma (MPM)
Description: FVC is the total amount of air exhaled during the Forced Expiratory Volume test. Baseline is defined as the most recent, non-missing value prior to or on the first study GSK3052230 treatment dose date. Change from Baseline is calculated as visit value minus Baseline value. Assessment of FVC was done on Day 1 of every odd cycle for Arm C participants with MPM. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates that data were not available as standard deviation could not be calculated for a single participant.
Time Frame: Up to 31 cycles (each cycle was of 21 days)
Population: All Treated Subjects Population
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
Number analyzed (Participants) | 3 | 25 | 8
Liters
  Cycle 3,Day 1, n=3, 24, 4: number analyzed (Participants) | 3 | 24 | 4
  Cycle 3,Day 1, n=3, 24, 4 | 0.303 (0.4688) | 0.280 (0.2911) | 0.138 (0.6762)
  Cycle 4,Day 1, n=1, 4, 1: number analyzed (Participants) | 1 | 4 | 1
  Cycle 4,Day 1, n=1, 4, 1 | -0.340 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant | 0.413 (0.1144) | 0.600 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant
  Cycle 5,Day 1, n=1, 23, 3: number analyzed (Participants) | 1 | 23 | 3
  Cycle 5,Day 1, n=1, 23, 3 | 0.240 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant | 0.238 (0.4178) | 0.587 (0.3592)
  Cycle 6,Day 1, n=1, 5, 2: number analyzed (Participants) | 1 | 5 | 2
  Cycle 6,Day 1, n=1, 5, 2 | 0.310 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant | 0.464 (0.3544) | 0.110 (0.8061)
  Cycle 7,Day 1, n=1, 15, 2: number analyzed (Participants) | 1 | 15 | 2
  Cycle 7,Day 1, n=1, 15, 2 | 0.530 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant | 0.399 (0.478) | 0.575 (0.0778)
  Cycle 8,Day 1, n=0, 3, 1: number analyzed (Participants) | 0 | 3 | 1
  Cycle 8,Day 1, n=0, 3, 1 |  | 0.263 (0.2371) | 0.640 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant
  Cycle 9,Day 1, n=0, 15, 1: number analyzed (Participants) | 0 | 15 | 1
  Cycle 9,Day 1, n=0, 15, 1 |  | 0.353 (0.4621) | 1.130 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant
  Cycle 10,Day 1, n=0, 3, 0: number analyzed (Participants) | 0 | 3 | 0
  Cycle 10,Day 1, n=0, 3, 0 |  | 0.063 (0.0751) |
  Cycle 11,Day 1, n=0, 12, 2: number analyzed (Participants) | 0 | 12 | 2
  Cycle 11,Day 1, n=0, 12, 2 |  | 0.347 (0.391) | 0.510 (0.6081)
  Cycle 12,Day 1, n=0, 2, 1: number analyzed (Participants) | 0 | 2 | 1
  Cycle 12,Day 1, n=0, 2, 1 |  | 0.225 (0.2333) | 0.580 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant
  Cycle 13,Day 1, n=0, 8, 2: number analyzed (Participants) | 0 | 8 | 2
  Cycle 13,Day 1, n=0, 8, 2 |  | 0.389 (0.42) | 0.555 (0.5162)
  Cycle 14,Day 1, n=0, 3, 1: number analyzed (Participants) | 0 | 3 | 1
  Cycle 14,Day 1, n=0, 3, 1 |  | -0.207 (0.65770) | 0.910 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant
  Cycle 15,Day 1, n=0, 6, 1: number analyzed (Participants) | 0 | 6 | 1
  Cycle 15,Day 1, n=0, 6, 1 |  | 0.247 (0.3406) | -0.030 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant
  Cycle 17,Day 1, n=0, 4, 1: number analyzed (Participants) | 0 | 4 | 1
  Cycle 17,Day 1, n=0, 4, 1 |  | 0.158 (0.3402) | 0.560 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant
  Cycle 19,Day 1, n=0, 1, 1: number analyzed (Participants) | 0 | 1 | 1
  Cycle 19,Day 1, n=0, 1, 1 |  | -0.02 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant | 0.620 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant
  Cycle 21,Day 1, n=0, 1, 1: number analyzed (Participants) | 0 | 1 | 1
  Cycle 21,Day 1, n=0, 1, 1 |  | -0.27 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant | 0.560 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant
  Cycle 23,Day 1, n=0, 1, 1: number analyzed (Participants) | 0 | 1 | 1
  Cycle 23,Day 1, n=0, 1, 1 |  | -0.62 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant | 0.510 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant
  Cycle 25,Day 1, n=0, 0, 1: number analyzed (Participants) | 0 | 0 | 1
  Cycle 25,Day 1, n=0, 0, 1 |  |  | 0.430 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant
  Cycle 27,Day 1, n=0, 0, 1: number analyzed (Participants) | 0 | 0 | 1
  Cycle 27,Day 1, n=0, 0, 1 |  |  | 0.220 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant
  Cycle 31,Day 1, n=0, 0, 1: number analyzed (Participants) | 0 | 0 | 1
  Cycle 31,Day 1, n=0, 0, 1 |  |  | 0.270 (NA) — NA indicates that data were not available as standard deviation could not be calculated for a single participant

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were be collected from the start of study treatment and up to Median of 28.5 weeks.
Description: All Treated Subjects Population
Arm/Group | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A | 5 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Docetaxel: Arm B | 20 mg/kg GSK3052230 + Docetaxel: Arm B | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/14 | 0/3 | 0/3 | 0/3 | 0/3 | 0/25 | 1/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/3 | 5/14 | 2/3 | 3/3 | 1/3 | 0/3 | 5/25 | 4/8
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 14/14 | 3/3 | 3/3 | 3/3 | 3/3 | 24/25 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A (N=3) | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A (N=3) | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A (N=14) | 5 mg/kg GSK3052230 + Docetaxel: Arm B (N=3) | 10 mg/kg GSK3052230 + Docetaxel: Arm B (N=3) | 20 mg/kg GSK3052230 + Docetaxel: Arm B (N=3) | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C (N=3) | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C (N=25) | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stenotrophomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A (N=3) | 10 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A (N=3) | 20 mg/kg GSK3052230 + Paclitaxel + Carboplatin: Arm A (N=14) | 5 mg/kg GSK3052230 + Docetaxel: Arm B (N=3) | 10 mg/kg GSK3052230 + Docetaxel: Arm B (N=3) | 20 mg/kg GSK3052230 + Docetaxel: Arm B (N=3) | 10 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C (N=3) | 15 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C (N=25) | 20 mg/kg GSK3052230 + Pemetrexed + Cisplatin: Arm C (N=8)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 1 (14) | 12 (50) | 1 (2) | 0 (0) | 2 (10) | 0 (0) | 6 (30) | 2 (6)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 5 (8) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (12) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (12) | 0 (0) | 0 (0) | 2 (10) | 0 (0) | 4 (12) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (4) | 2 (8) | 3 (13) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 6 (29) | 3 (16)
Fatigue (General disorders) | 0 (0) | 1 (1) | 5 (12) | 2 (2) | 1 (1) | 1 (3) | 1 (1) | 10 (11) | 5 (6)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 6 (7) | 2 (6)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Dysaesthesia (Nervous system disorders) | 3 (4) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Neurotoxicity (Nervous system disorders) | 1 (1) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Peripheral sensory neuropathy (General disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Dysgeusia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 2 (2)
Syncope (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (4) | 2 (2) | 7 (8) | 2 (6) | 0 (0) | 1 (1) | 2 (2) | 3 (5) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (3) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 7 (9) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (4) | 3 (5) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 12 (27) | 7 (20)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (9) | 5 (14)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (3) | 4 (6) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 7 (9) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 3 (3) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 8 (10) | 5 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 5 (11) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (7) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (6) | 2 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (10) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 2 (4) | 1 (6) | 2 (4) | 5 (18) | 1 (6)
Blood creatinine increased (Investigations) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 5 (12) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (11) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (6) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 7 (10) | 4 (6)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystoid macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal neovascularisation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymph node palpable (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (4) | 1 (2)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (8) | 0 (0)
Thrombosis in device (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (8) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Salivary duct inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood fibrinogen increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram repolarisation abnormality (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT01868022/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT01868022/SAP_001.pdf